CLINICAL TRIAL: NCT00047333
Title: A Phase 2 Open-Label Study Of OSI-774 (NSC 718781) In Unresectable Hepatocellular Carcinoma
Brief Title: Erlotinib in Treating Patients With Liver Cancer That Cannot be Surgically Removed
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Administratively complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02498; ID02-008; CDR0000257665 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2002-10-03; First posted 2003-01-27 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Adult Primary Hepatocellular Carcinoma; Advanced Adult Primary Liver Cancer; Localized Unresectable Adult Primary Liver Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Erlotinib Hydrochloride

ARMS (1):
- Treatment (erlotinib hydrochloride) (Experimental): Patients receive oral erlotinib once daily. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: erlotinib hydrochloride; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: erlotinib hydrochloride — Given PO
  Other Names: CP-358,774; erlotinib; OSI-774
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
Phase II trial to study the effectiveness of erlotinib in treating patients who have liver cancer that cannot be surgically removed. Erlotinib may stop the growth of tumor cells by blocking the enzymes necessary for their growth

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess progression-free survival (PFS) measured at 16 weeks following initiation of once daily continuous oral therapy with OSI-774 in patients with unresectable hepatocellular carcinoma.

SECONDARY OBJECTIVES:

I. To assess objective response rate, rate and duration of stable disease, time to progression, median and overall survival in this patient population, and any changes in tumor perfusion based on functional CT imaging.

II. To correlate response with patient characteristics including: age, disease stage (TNM, Okuda [6]), viral hepatitis status, pathologic grade of cirrhosis, Childs-Pugh status, Performance Status, serum values of: alpha feto-protein, bilirubin, transaminases, albumin; EGFR expression score by IHC; and development of skin rash during therapy.

III. To determine the pharmacokinetic and pharmacodynamic profile of OSI-774 in this patient population.

IV. To determine the safety and tolerability of OSI-774 in this patient population.

OUTLINE: Patients are stratified according to epidermal growth factor receptor expression (low, 0-1+ vs high, 2-3+).

Patients receive oral erlotinib once daily. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed hepatocellular carcinoma (HCC)not amenable to curative resection

  * No fibrolamellar HCC
* No prior therapy for HCC, including systemic chemotherapy, hepatic arterial infusion of chemotherapeutic agents or irradiated microspheres, and epidermal growth factor receptor-targeting agents

  * The following prior therapies are allowed provided previously treated lesions remain separate from those to be evaluated in present study

    * Surgery
    * Liver-directed therapy (e.g., radiofrequency ablation, transarterial embolization/chemoembolization, or percutaneous ethanol injection)
* At least 1 unidimensionally measurable lesion

  * At least 20 mm by conventional techniques
* Must have paraffin tissue block or unstained slides from biopsy or surgical specimen
* No known brain metastases
* No ascites that are refractory to conservative management (e.g., sodium restriction to 50 mEq/day dietary sodium and fluid restrictions and/or diuretics)
* Performance status - ECOG 0-2
* At least 16 weeks
* Granulocyte count at least 1,500/mm^3
* Platelet count at least 60,000/mm^3
* Hemoglobin at least 10 g/dL
* Bilirubin no greater than 1.8 mg/dL
* Albumin at least 2.5 g/dL
* AST/ALT no greater than 5 times upper limit of normal
* PT no greater than 1-3 seconds over normal
* No decompensated liver disease
* No jaundice
* No portosystemic encephalopathy (evidenced by confusion, asterixis, significant sleep disturbance, or hypothermia less than 36º Celsius)
* No hyponatremia with sodium less than 125 mEq/L
* No portal hypertension with bleeding esophageal or gastric varices within the past 3 months
* Creatinine no greater than 2 mg/dL
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No gastrointestinal tract disease resulting in an inability to take oral medication or requirement for IV alimentation
* No active peptic ulcer disease
* No abnormalities of the cornea (e.g., dry eye syndrome or Sjögren's syndrome)
* No congenital abnormality (e.g., Fuch's dystrophy)
* No other uncontrolled concurrent illness that would preclude study participation
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No other malignancy within the past 5 years except nonmelanoma skin cancer
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior surgical therapy affecting absorption
* More than 30 days since prior investigational agents
* No concurrent commercial or other investigational anticancer agents or therapies
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2002-08; Primary Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | Time from initiation of therapy until documented disease progression, assessed at 16 weeks
  Summarized by Kaplan-Meier curves, from which medians and progression-free survival can be attained.

SECONDARY OUTCOMES:
Objective response rate | Up to 4 years
  Summarized by estimates and standard errors.
Rate of stable disease | Up to 4 years
  Summarized by estimates and standard errors.
Duration of stable disease | From the start of the treatment until the criteria for progression are met, assessed up to 4 years
  Summarized by Kaplan-Meier curves, from which medians and overall duration of stable disease can be attained.
Time to progression | Up to 4 years
  Summarized by Kaplan-Meier curves, from which medians and time to progression can be attained.
Overall survival | Up to 4 years
  Summarized by Kaplan-Meier curves, from which medians and overall survival can be attained.

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Thomas, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States